CLINICAL TRIAL: NCT01991457
Title: Single Arm Phase II Study of Myeloablative Allogeneic Hematopoietic Stem Cell Transplantation for Acute Lymphoblastic Leukemia (ALL) in Older Patients Using Fludarabine and Total Body Irradiation (FluTBI) Regimen
Brief Title: Fludarabine / Total Body Irradiation Regimen for ALLO HCT in Acute Lymphoblastic Leukemia
Acronym: FluTBI
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Omer Jamy, Primary Investigator, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UAB 1285
Record Dates: First submitted 2013-09-29; First posted 2013-11-25 (Estimated); Results first posted 2022-09-21 (Actual); Last update posted 2024-01-12 (Actual); Status verified 2024-01

CONDITIONS: Adult Lymphoblastic Lymphoma
Keywords: ALL
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — fludarabine; Whole-Body Irradiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes

ARMS (1):
- Treatment (Other): Fludarabine, Total Body Irradiation (TBI) Fludarabine: 40 mg/m2 X 4 days TBI: TBI 2 Gy 2 times a day X 3 days
  Interventions: Drug: Fludarabine; Procedure: Total Body Irradiation

INTERVENTIONS:
Drug: Fludarabine
Procedure: Total Body Irradiation

SUMMARY:
The goal of this research is to test if the conditioning regimen, fludarabine and total body irradiation (FluTBI), can lead to a safer and more effective stem cell transplant treatment regimen for ALL patients older than 40 years of age and/or younger patients with high risk medical conditions. The primary objective is to establish the efficacy of allo HCT in older ALL patients using myeloablative FluTBI conditioning regimen. The investigators are also assessing the safety and toxicity of allo HCT in older ALL patients using myeloablative FluTBI conditioning regimen.

ELIGIBILITY:
Inclusion Criteria:

* Disease Criteria:

  * ALL in complete remission (CR) at the time of transplant. Remission is defined as "less than 5.0% bone marrow lymphoblasts by morphology," as determined by a bone marrow aspirate obtained within 2 weeks of study registration.
  * Philadelphia chromosome positive ALL is allowed.
  * Lymphoid blastic crisis of CML will be included (provided that patients achieve CR).
* Age Criteria: Equal or above age 40 and up to 65 years. If younger than 40, there must be comorbidities which preclude the patient to undergo CyTBI conditioning regimen.
* Organ Function Criteria: All organ function testing should be done within 28 days of study registration.
* Cardiac: Left ventricular ejection fraction (LVEF) ≥ 50% by MUGA (Multi Gated Acquisition) scan or echocardiogram.
* Pulmonary: FEV1 (Forced expiratory volume in 1 second) and FVC (Forced vital capacity) ≥ 50% predicted, DLCO (alveolar diffusion capacity for carbon monoxide) (corrected for hemoglobin) ≥ 50% of predicted.
* Renal: The estimated creatinine clearance (CrCl) must be equal or greater than 60 mL/min/1.73 m2 as calculated by the Cockcroft-Gault Formula:

CrCl = (140-age) x weight (kg) x 0.85 (if female)/72 x serum creatinine (mg/dL).

* Hepatic:

  * Serum bilirubin 2.0 g/dL
  * Aspartate transaminase (AST)/alanine transaminase (ALT) 2.5 ULN
  * Alkaline phosphatase 2.5 ULN
* Performance status: Karnofsky ≥ 70%
* Consent: Patient must be informed of the investigational nature of this study in accordance with institutional and federal guidelines and have the ability to provide written informed consent prior to initiation of any study-related procedures, and ability,in the opinion of the principal investigator, to comply with all the requirements of the study.
* Presence of a willing adult HLA-matched sibling (excluding identical twin) or HLA-matched unrelated donor meeting all the criteria for routine allo HSCT. All donors will be evaluated for eligibility and suitability per the standard of care according to the FACT and NMDP guidelines.

Exclusion Criteria:

* Non-compliant to medications.
* No appropriate caregivers identified.
* HIV1 (Human Immunodeficiency Virus-1) or HIV2 positive
* Active life-threatening cancer requiring treatment other than ALL
* Uncontrolled medical or psychiatric disorders.
* Uncontrolled infections, defined as positive blood cultures within 72 hours of study entry, or evidence of progressive infection by imaging studies such as chest CT scan within 14 days of registration.
* Active central nervous system (CNS) leukemia
* Preceding allogeneic HSCT
* Receiving intensive chemotherapy within 21 days of registration. Maintenance type of chemotherapy will be allowed.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2013-08-27 (Actual); Primary Completion 2020-01-30 (Actual); Study Completion 2022-08-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Omer H Jamy, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- UAB Bone Marrow Transplantation and Cellular Therapy Program, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gaynon PS, Angiolillo AL, Carroll WL, Nachman JB, Trigg ME, Sather HN, Hunger SP, Devidas M; Children's Oncology Group. Long-term results of the children's cancer group studies for childhood acute lymphoblastic leukemia 1983-2002: a Children's Oncology Group Report. Leukemia. 2010 Feb;24(2):285-97. doi: 10.1038/leu.2009.262. Epub 2009 Dec 17. PMID 20016531
- [Background] Annino L, Vegna ML, Camera A, Specchia G, Visani G, Fioritoni G, Ferrara F, Peta A, Ciolli S, Deplano W, Fabbiano F, Sica S, Di Raimondo F, Cascavilla N, Tabilio A, Leoni P, Invernizzi R, Baccarani M, Rotoli B, Amadori S, Mandelli F; GIMEMA Group. Treatment of adult acute lymphoblastic leukemia (ALL): long-term follow-up of the GIMEMA ALL 0288 randomized study. Blood. 2002 Feb 1;99(3):863-71. doi: 10.1182/blood.v99.3.863. PMID 11806988
- [Background] Alvarnas JC, Brown PA, Aoun P, Ballen KK, Bellam N, Blum W, Boyer MW, Carraway HE, Coccia PF, Coutre SE, Cultrera J, Damon LE, DeAngelo DJ, Douer D, Frangoul H, Frankfurt O, Goorha S, Millenson MM, O'Brien S, Petersdorf SH, Rao AV, Terezakis S, Uy G, Wetzler M, Zelenetz AD, Naganuma M, Gregory KM; National Comprehensive Cancer Network. Acute lymphoblastic leukemia. J Natl Compr Canc Netw. 2012 Jul 1;10(7):858-914. doi: 10.6004/jnccn.2012.0089. PMID 22773801
- [Background] Larson RA, Dodge RK, Burns CP, Lee EJ, Stone RM, Schulman P, Duggan D, Davey FR, Sobol RE, Frankel SR, et al. A five-drug remission induction regimen with intensive consolidation for adults with acute lymphoblastic leukemia: cancer and leukemia group B study 8811. Blood. 1995 Apr 15;85(8):2025-37. PMID 7718875
- [Background] Yanada M, Matsuo K, Suzuki T, Naoe T. Allogeneic hematopoietic stem cell transplantation as part of postremission therapy improves survival for adult patients with high-risk acute lymphoblastic leukemia: a metaanalysis. Cancer. 2006 Jun 15;106(12):2657-63. doi: 10.1002/cncr.21932. PMID 16703597
- [Background] Bachanova V, Weisdorf D. Unrelated donor allogeneic transplantation for adult acute lymphoblastic leukemia: a review. Bone Marrow Transplant. 2008 Mar;41(5):455-64. doi: 10.1038/sj.bmt.1705889. Epub 2007 Oct 29. PMID 17968329
- [Background] Hahn T, Wall D, Camitta B, Davies S, Dillon H, Gaynon P, Larson RA, Parsons S, Seidenfeld J, Weisdorf D, McCarthy PL Jr. The role of cytotoxic therapy with hematopoietic stem cell transplantation in the therapy of acute lymphoblastic leukemia in adults: an evidence-based review. Biol Blood Marrow Transplant. 2006 Jan;12(1):1-30. doi: 10.1016/j.bbmt.2005.10.018. PMID 16399566
- [Background] Chaidos A, Kanfer E, Apperley JF. Risk assessment in haemotopoietic stem cell transplantation: disease and disease stage. Best Pract Res Clin Haematol. 2007 Jun;20(2):125-54. doi: 10.1016/j.beha.2006.10.003. PMID 17448953
- [Background] Goldstone AH, Richards SM, Lazarus HM, Tallman MS, Buck G, Fielding AK, Burnett AK, Chopra R, Wiernik PH, Foroni L, Paietta E, Litzow MR, Marks DI, Durrant J, McMillan A, Franklin IM, Luger S, Ciobanu N, Rowe JM. In adults with standard-risk acute lymphoblastic leukemia, the greatest benefit is achieved from a matched sibling allogeneic transplantation in first complete remission, and an autologous transplantation is less effective than conventional consolidation/maintenance chemotherapy in all patients: final results of the International ALL Trial (MRC UKALL XII/ECOG E2993). Blood. 2008 Feb 15;111(4):1827-33. doi: 10.1182/blood-2007-10-116582. Epub 2007 Nov 29. PMID 18048644
- [Background] Ringden O, Labopin M, Tura S, Arcese W, Iriondo A, Zittoun R, Sierra J, Gorin NC. A comparison of busulphan versus total body irradiation combined with cyclophosphamide as conditioning for autograft or allograft bone marrow transplantation in patients with acute leukaemia. Acute Leukaemia Working Party of the European Group for Blood and Marrow Transplantation (EBMT). Br J Haematol. 1996 Jun;93(3):637-45. doi: 10.1046/j.1365-2141.1996.d01-1681.x. PMID 8652385
- [Background] Davies SM, Ramsay NK, Klein JP, Weisdorf DJ, Bolwell B, Cahn JY, Camitta BM, Gale RP, Giralt S, Heilmann C, Henslee-Downey PJ, Herzig RH, Hutchinson R, Keating A, Lazarus HM, Milone GA, Neudorf S, Perez WS, Powles RL, Prentice HG, Schiller G, Socie G, Vowels M, Wiley J, Yeager A, Horowitz MM. Comparison of preparative regimens in transplants for children with acute lymphoblastic leukemia. J Clin Oncol. 2000 Jan;18(2):340-7. doi: 10.1200/JCO.2000.18.2.340. PMID 10637248
- [Background] Marks DI, Forman SJ, Blume KG, Perez WS, Weisdorf DJ, Keating A, Gale RP, Cairo MS, Copelan EA, Horan JT, Lazarus HM, Litzow MR, McCarthy PL, Schultz KR, Smith DD, Trigg ME, Zhang MJ, Horowitz MM. A comparison of cyclophosphamide and total body irradiation with etoposide and total body irradiation as conditioning regimens for patients undergoing sibling allografting for acute lymphoblastic leukemia in first or second complete remission. Biol Blood Marrow Transplant. 2006 Apr;12(4):438-53. doi: 10.1016/j.bbmt.2005.12.029. PMID 16545728
- [Background] Snyder DS, Nademanee AP, O'Donnell MR, Parker PM, Stein AS, Margolin K, Somlo G, Molina A, Spielberger R, Kashyap A, Fung H, Slovak ML, Dagis A, Negrin RS, Amylon MD, Blume KG, Forman SJ. Long-term follow-up of 23 patients with Philadelphia chromosome-positive acute lymphoblastic leukemia treated with allogeneic bone marrow transplant in first complete remission. Leukemia. 1999 Dec;13(12):2053-8. doi: 10.1038/sj.leu.2401589. PMID 10602428
- [Background] Horowitz MM, Gale RP, Sondel PM, Goldman JM, Kersey J, Kolb HJ, Rimm AA, Ringden O, Rozman C, Speck B, et al. Graft-versus-leukemia reactions after bone marrow transplantation. Blood. 1990 Feb 1;75(3):555-62. PMID 2297567
- [Background] Gale RP, Horowitz MM. Graft-versus-leukemia in bone marrow transplantation. The Advisory Committee of the International Bone Marrow Transplant Registry. Bone Marrow Transplant. 1990 Jul;6 Suppl 1:94-7. PMID 2390646
- [Background] Arnold R, Massenkeil G, Bornhauser M, Ehninger G, Beelen DW, Fauser AA, Hegenbart U, Hertenstein B, Ho AD, Knauf W, Kolb HJ, Kolbe K, Sayer HG, Schwerdtfeger R, Wandt H, Hoelzer D. Nonmyeloablative stem cell transplantation in adults with high-risk ALL may be effective in early but not in advanced disease. Leukemia. 2002 Dec;16(12):2423-8. doi: 10.1038/sj.leu.2402712. PMID 12454748
- [Background] Martino R, Giralt S, Caballero MD, Mackinnon S, Corradini P, Fernandez-Aviles F, San Miguel J, Sierra J. Allogeneic hematopoietic stem cell transplantation with reduced-intensity conditioning in acute lymphoblastic leukemia: a feasibility study. Haematologica. 2003 May;88(5):555-60. PMID 12745275
- [Background] Hamaki T, Kami M, Kanda Y, Yuji K, Inamoto Y, Kishi Y, Nakai K, Nakayama I, Murashige N, Abe Y, Ueda Y, Hino M, Inoue T, Ago H, Hidaka M, Hayashi T, Yamane T, Uoshima N, Miyakoshi S, Taniguchi S. Reduced-intensity stem-cell transplantation for adult acute lymphoblastic leukemia: a retrospective study of 33 patients. Bone Marrow Transplant. 2005 Mar;35(6):549-56. doi: 10.1038/sj.bmt.1704776. PMID 15756282
- [Background] Gutierrez-Aguirre CH, Gomez-Almaguer D, Cantu-Rodriguez OG, Gonzalez-Llano O, Jaime-Perez JC, Herena-Perez S, Manzano CA, Estrada-Gomez R, Gonzalez-Carrillo ML, Ruiz-Arguelles GJ. Non-myeloablative stem cell transplantation in patients with relapsed acute lymphoblastic leukemia: results of a multicenter study. Bone Marrow Transplant. 2007 Sep;40(6):535-9. doi: 10.1038/sj.bmt.1705769. Epub 2007 Jul 9. PMID 17618317
- [Background] Mohty M, Labopin M, Tabrizzi R, Theorin N, Fauser AA, Rambaldi A, Maertens J, Slavin S, Majolino I, Nagler A, Blaise D, Rocha V; Acute Leukemia Working Party; European Group for Blood and Marrow Transplantation. Reduced intensity conditioning allogeneic stem cell transplantation for adult patients with acute lymphoblastic leukemia: a retrospective study from the European Group for Blood and Marrow Transplantation. Haematologica. 2008 Feb;93(2):303-6. doi: 10.3324/haematol.11960. PMID 18245655
- [Background] Devine SM, Sanborn R, Jessop E, Stock W, Huml M, Peace D, Wickrema A, Yassine M, Amin K, Thomason D, Chen YH, Devine H, Maningo M, van Besien K. Fludarabine and melphalan-based conditioning for patients with advanced hematological malignancies relapsing after a previous hematopoietic stem cell transplant. Bone Marrow Transplant. 2001 Sep;28(6):557-62. doi: 10.1038/sj.bmt.1703198. PMID 11607768
- [Background] Ciurea SO, Saliba RM, Hamerschlak N, Karduss Aurueta AJ, Bassett R, Fernandez-Vina M, Petropoulos D, Worth LL, Chan KW, Couriel DR, Rondon G, Sharma M, Qazilbash M, Jones RB, Kebriaei P, McMannis J, Hosing CM, Nieto Y, Champlin RE, Shpall EJ, de Lima M. Fludarabine, melphalan, thiotepa and anti-thymocyte globulin conditioning for unrelated cord blood transplant. Leuk Lymphoma. 2012 May;53(5):901-6. doi: 10.3109/10428194.2011.631159. Epub 2012 Jan 3. PMID 21988645
- [Background] Ram R, Storb R, Sandmaier BM, Maloney DG, Woolfrey A, Flowers ME, Maris MB, Laport GG, Chauncey TR, Lange T, Langston AA, Storer B, Georges GE. Non-myeloablative conditioning with allogeneic hematopoietic cell transplantation for the treatment of high-risk acute lymphoblastic leukemia. Haematologica. 2011 Aug;96(8):1113-20. doi: 10.3324/haematol.2011.040261. Epub 2011 Apr 20. PMID 21508120
- [Background] Alousi A, de Lima M. Reduced-intensity conditioning allogeneic hematopoietic stem cell transplantation. Clin Adv Hematol Oncol. 2007 Jul;5(7):560-70. PMID 17679930
- [Background] Kroger N, Bornhauser M, Ehninger G, Schwerdtfeger R, Biersack H, Sayer HG, Wandt H, Schafer-Eckardt K, Beyer J, Kiehl M, Zander AR; German Cooperative Transplant Study Group. Allogeneic stem cell transplantation after a fludarabine/busulfan-based reduced-intensity conditioning in patients with myelodysplastic syndrome or secondary acute myeloid leukemia. Ann Hematol. 2003 Jun;82(6):336-42. doi: 10.1007/s00277-003-0654-9. Epub 2003 May 1. PMID 12728337
- [Background] Stelljes M, Bornhauser M, Kroger M, Beyer J, Sauerland MC, Heinecke A, Berning B, Scheffold C, Silling G, Buchner T, Neubauer A, Fauser AA, Ehninger G, Berdel WE, Kienast J; Cooperative German Transplant Study Group. Conditioning with 8-Gy total body irradiation and fludarabine for allogeneic hematopoietic stem cell transplantation in acute myeloid leukemia. Blood. 2005 Nov 1;106(9):3314-21. doi: 10.1182/blood-2005-04-1377. Epub 2005 Jul 14. PMID 16020510
- [Background] Nakamura Y, Mori T, Kato J, Aisa Y, Nakazato T, Shigematsu N, Okamoto S. [Allogeneic hematopoietic stem cell transplantation with fludarabine, melphalan, and total body irradiation as a conditioning for elderly patients with myeloid malignancies]. Rinsho Ketsueki. 2012 Mar;53(3):318-22. Japanese. PMID 22499048
- [Background] Przepiorka D, Weisdorf D, Martin P, Klingemann HG, Beatty P, Hows J, Thomas ED. 1994 Consensus Conference on Acute GVHD Grading. Bone Marrow Transplant. 1995 Jun;15(6):825-8. PMID 7581076
- [Background] Fiere D, Lepage E, Sebban C, Boucheix C, Gisselbrecht C, Vernant JP, Varet B, Broustet A, Cahn JY, Rigal-Huguet F, et al. Adult acute lymphoblastic leukemia: a multicentric randomized trial testing bone marrow transplantation as postremission therapy. The French Group on Therapy for Adult Acute Lymphoblastic Leukemia. J Clin Oncol. 1993 Oct;11(10):1990-2001. doi: 10.1200/JCO.1993.11.10.1990. PMID 8410124
- [Background] Sebban C, Lepage E, Vernant JP, Gluckman E, Attal M, Reiffers J, Sutton L, Racadot E, Michallet M, Maraninchi D, et al. Allogeneic bone marrow transplantation in adult acute lymphoblastic leukemia in first complete remission: a comparative study. French Group of Therapy of Adult Acute Lymphoblastic Leukemia. J Clin Oncol. 1994 Dec;12(12):2580-7. doi: 10.1200/JCO.1994.12.12.2580. PMID 7989932
- See also: UAB Bone Marrow Transplantation and Cell Therapy Program — http://www.uab.edu/medicine/bonemarrow/

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment: Fludarabine, Total Body Irradiation (TBI)
  Fludarabine
  Total Body Irradiation
Period: Overall Study
Arm/Group | Treatment
Started | 19
Completed | 19
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment
Number analyzed (Participants) | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 19
  >=65 years | 0
Age, Continuous [Median (Full Range); unit: years] | 54 [44 to 63]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 10
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Non-Hispanic White | 19
Region of Enrollment [Number; unit: participants]
  United States | 19

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects Disease-free Survival
Description: Percentage of patients without relapse of disease at 2 years
Time Frame: 2 years post-transplant
Measure: Number; unit: percentage of participants
Arm/Group | Treatment
Number analyzed (Participants) | 19
percentage of participants | 63.2

2. Secondary Outcome: Percentage of Subjects That Survived
Time Frame: 2 years post-transplant
Measure: Number; unit: Percentage of subjects that survived
Groups:
- Treatment: Fludarabine, Total Body Irradiation (TBI) Fludarabine: 40 mg/m2 X 4 days TBI: TBI 2 Gy 2 times a day X 3 days
  Fludarabine
  Total Body Irradiation
Arm/Group | Treatment
Number analyzed (Participants) | 19
Percentage of subjects that survived | 68.4

3. Secondary Outcome: Time to Neutrophil Engraftment
Description: Neutrophil engraftment is defined as the first of 3 consecutive days with an absolute neutrophil count (ANC) > 500/μL. Measuring the number of days it takes for (ANC) > 500/μL.
Time Frame: Within the first 100 days
Measure: Median (Full Range); unit: days
Arm/Group | Treatment
Number analyzed (Participants) | 19
days | 12 [10 to 24]

4. Secondary Outcome: Number of Subjects With Regimen Related Toxicity
Time Frame: Within first 100 days post-transplant
Measure: Number; unit: participants
Arm/Group | Treatment
Number analyzed (Participants) | 19
participants
  Acute kidney injury* | 4
  Gastrointestinal (GI | 4
  Mucositis | 3

5. Secondary Outcome: Percentage of Subjects With Acute GVHD
Time Frame: 2 years post transplant
Measure: Number; unit: percentage of aGVHD
Arm/Group | Treatment
Number analyzed (Participants) | 19
percentage of aGVHD | 26.1

6. Secondary Outcome: Number of Patients With Immune Reconstitution
Time Frame: 1 year post transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment
Number analyzed (Participants) | 19
Participants | 19

7. Secondary Outcome: Percentage of Subjects With Relapse
Time Frame: 2 Years post-transplant
Measure: Number; unit: percentage of subjects with relapse
Arm/Group | Treatment
Number analyzed (Participants) | 19
percentage of subjects with relapse | 7.1

8. Secondary Outcome: Number of Subjects With Platelet Engraftment
Description: Platelet engraftment is defined as the first of 3 consecutive days with a platelet count > 20,000/μL without platelet transfusion for 7 days.
Time Frame: Within 100 days post transplant
Measure: Number; unit: Number of subjects with platelet engraft
Arm/Group | Treatment
Number analyzed (Participants) | 19
Number of subjects with platelet engraft | 19

9. Secondary Outcome: Percentage of Subjects With Chronic GVHD
Time Frame: 2 years post transplant
Measure: Number; unit: Percentage of subjects with chronic GVHD
Arm/Group | Treatment
Number analyzed (Participants) | 19
Percentage of subjects with chronic GVHD | 32

ADVERSE EVENTS:
Time Frame: 100 days
Arm/Group | Treatment
All-Cause Mortality (participants affected / at risk) | 3/19
Serious Adverse Events (participants affected / at risk) | 11/19
Other Adverse Events (participants affected / at risk) | 5/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (N=19)
Acute kidney injury (Renal and urinary disorders) | 4
Gastrointestinal (GI) (Gastrointestinal disorders) | 4
Mucositis (Gastrointestinal disorders) | 3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (N=19)
Atrial flutter (Cardiac disorders) | 1
Encephalopathy (Nervous system disorders) | 1
Hyponatremia (Renal and urinary disorders) | 1
Elevated liver enzymes (Hepatobiliary disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-12-09): https://cdn.clinicaltrials.gov/large-docs/57/NCT01991457/Prot_SAP_002.pdf
  • Informed Consent Form (2018-12-09): https://cdn.clinicaltrials.gov/large-docs/57/NCT01991457/ICF_003.pdf